CLINICAL TRIAL: NCT03854032
Title: Window-of-Opportunity Trial of Nivolumab and BMS986205 in Patients With Squamous Cell Carcinoma of the Head and Neck (CA017-087)
Brief Title: Nivolumab and BMS986205 in Treating Patients With Stage II-IV Squamous Cell Cancer of the Head and Neck
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18P.771; JT 13241 (Other: JeffTrial Number)
Record Dates: First submitted 2019-02-21; First posted 2019-02-26 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Lip; Oral Cavity Squamous Cell Carcinoma; Pharynx; Larynx; Squamous Cell Carcinoma
MeSH Terms: conditions — Lymphoid Interstitial Pneumonia; Squamous Cell Carcinoma of Head and Neck; Laryngeal Diseases; Carcinoma, Squamous Cell | interventions — Nivolumab; linrodostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (BMS986205, nivolumab) (Experimental): Patients receive IDO1 inhibitor BMS-986205 PO QD. Beginning week 2, patients also receive nivolumab IV over 30 minutes on day 1. Treatment repeats for up to 5 weeks in the absence of disease progression or unacceptable toxicity. Patients showing a treatment response receive IDO1 inhibitor BMS-986205 PO QD for 4 additional weeks and receive nivolumab IV over 30 minutes on day 1, then undergo surgery at week 10. Those without a treatment response after 5 weeks undergo surgery within 7 days.
  Interventions: Biological: Nivolumab; Biological: IDO1 Inhibitor BMS-986205; Procedure: Therapeutic Conventional Surgery; Other: Questionnaire Administration
- Arm II (nivolumab) (Active Comparator): Patients receive nivolumab IV over 30 minutes on day 1 in the absence of disease progression or unacceptable toxicity. Patients showing treatment response after 4 weeks receive nivolumab IV over 30 minutes on day 1, then undergo surgery at week 9. Those without a treatment response after 4 weeks undergo surgery within 7 days.
  Interventions: Biological: Nivolumab; Procedure: Therapeutic Conventional Surgery; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Nivolumab — Given IV
  Other Names: 946414-94-4; BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Biological: IDO1 Inhibitor BMS-986205 — Given PO
  Other Names: (R)-N-(4-chlorophenyl)-2-((1S,4S)-4-(6-fluoroquinolin-4-yl)cyclohexyl)propenamide; BMS 986205; BMS-986205; BMS986205; IDO-1 Inhibitor BMS-986205; Indoleamine-pyrrole 2,3-Dioxygenase Inhibitor BMS-986205; ONO-7701
  Arms: Arm I (BMS986205, nivolumab)
Procedure: Therapeutic Conventional Surgery — Undergo Surgery
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well nivolumab works, with or without BMS986205, in treating patients with stage II-IV squamous cell cancer of the head and neck. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. BMS986205 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving nivolumab with BMS986205 may work better than nivolumab alone in treating patients with squamous cell cancer of the head and neck.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the impact of IDO1 inhibitor BMS-986205 (BMS986205) and nivolumab versus nivolumab alone on tumor radiographic response both at the primary tumor site and in regional lymph nodes by investigator assessment at 5 weeks.

SECONDARY OBJECTIVES:

I. To investigate whether adding the IDO1 - inhibitor, BMS986205, to nivolumab therapy affects intratumoral and systemic anti-tumor immunity.

II. To assess the impact of BMS986205 and nivolumab verses nivolumab alone on pathologic treatment effect bother at the primary and regional lymph nodes.

III. To determine the effect of BMS986205 and nivolumab versus nivolumab alone on immune cell composition within the tumor microenvironment including the presence of effector T cells (Teff), regulatory T cells (Treg), and tumor-associated macrophages (TAM).

IV. To further characterize the effect of BMS986205 when combined with nivolumab on kynurenine production and correlate these levels with effects on immune cell composition and polarization.

V. To review the relationship of p16 status by immunohistochemistry with immune cell polarization, tumor radiographic response, and immune cell composition.

VI. To review the relationship of PD-L1 status by immunohistochemistry with immune cell polarization, tumor radiographic response, and immune cell composition.

VII. To assess the safety and tolerability of BMS986205 and nivolumab. VIII. Evaluate surgical wound healing post treatment.

EXPLORATORY OBJECTIVES:

I. To further characterize the effect of BMS986205 and nivolumab versus nivolumab alone through analysis of T cell repertoire.

II. To assess the interactions between the immune and metabolic microenvironment through analysis of alterations in exosome composition in peripheral blood as it related to immune, cytokine and metabolic alterations before, during and after treatment.

III. To identify risks for poor physical and mental health outcomes; examine bio-behavioral factors associated with cancer treatment outcomes; and evaluate the physical and psychosocial needs of cancer survivors through patient reported outcomes.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive IDO1 inhibitor BMS-986205 orally (PO) once daily (QD). Beginning week 2, patients also receive nivolumab intravenously (IV) over 30 minutes on day 1. Treatment repeats for up to 5 weeks in the absence of disease progression or unacceptable toxicity. Patients showing a treatment response receive IDO1 inhibitor BMS-986205 PO QD for 4 additional weeks and receive nivolumab IV over 30 minutes on day 1, then undergo surgery at week 10. Those without a treatment response after 5 weeks undergo surgery within 7 days.

ARM II: Patients receive nivolumab IV over 30 minutes on day 1 in the absence of disease progression or unacceptable toxicity. Patients showing treatment response after 4 weeks receive nivolumab IV over 30 minutes on day 1, then undergo surgery at week 9. Those without a treatment response after 4 weeks undergo surgery within 7 days.

After completion of study treatment, patients are followed up periodically for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed head and neck squamous cell carcinoma (HNSC).
* Any stage 2 or greater HNSCC (American Joint Committee on Cancer [AJCC] 8th edition) of the 1) oral cavity, 2) larynx, 3) hypopharynx, 4) nasal cavity/paranasal sinuses or 5) stage 1 oropharyngeal with lymphadenopathy. Patients with resectable disease that is amenable to surgery are eligible. Patient must have been determined to be candidates for surgical resection by a multi-disciplinary team including a surgeon, a medical oncologist
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* White blood cells 2000/ul or more.
* Absolute neutrophil count 1500/ul or more.
* Platelets 100,000/ul or more.
* Hemoglobin 9 g/dl or more.
* Bilirubin less than or equal to 1.5 x the upper limit of normal (except subjects with Gilbert syndrome, who can have total bilirubin < 3 mg/dl).
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3 x the upper limit of normal.
* Glomerular filtration rate (GFR) greater than or equal to 40 ml/min using the Cockcroft-Gault formula or serum creatinine less than or equal to 1.5 x ULN.
* Women of child bearing potential (WOCBP) should have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 21 days of study enrollment.
* WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study treatment(s) plus 5 months post-treatment completion.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study treatment(s) plus 7 months post-treatment completion. In addition, male participants must be willing to refrain from sperm donation during this time.
* Males who are sexually active with WOCBP must agree to use a condom during any sexual activity for the duration of treatment with study treatment plus 7 months after the last dose of the study treatment (i.e., 90 days [duration of sperm turnover] plus the time required for nivolumab to undergo approximately 5 half-lives). This criterion applies to azoospermic males as well. In addition, male participants must be willing to refrain from sperm donation during this time.

  * Male mandatory condom use is regardless of whether the participant has undergone a successful vasectomy or if the female partner is pregnant.
  * Investigators shall counsel WOCBP, and male participants who are sexually active with WOCBP, on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise on the use of highly effective methods of contraception, which have a failure rate of < 1% when used consistently and correctly. Hormonal contraceptives are prohibited methods of contraception for participants receiving BMS-986205 this study who are WOCBP.
* All subjects must be able to comprehend and sign a written informed consent document.

Exclusion Criteria:

* Patients with nasopharyngeal carcinoma, salivary gland or skin primaries.
* Patients with recurrent head and neck cancer treated previously with chemotherapy, radiation or immunotherapy.
* Any history of a severe hypersensitivity reaction to any monoclonal antibody.
* Any history of allergy to the study drug components.
* Participants with a personal or family (i.e., in a first-degree relative) history or presence of cytochrome b5 reductase deficiency (previously called methemoglobin reductase deficiency) or other diseases that puts them at risk of methemoglobinemia. All participants will be screened for methemoglobin levels prior to randomization.
* Participants with a history of G6PD deficiency or other congenital or autoimmune hemolytic disorders. All participants will be screened for G6PD deficiency prior to randomization.
* Participants with history of serotonin syndrome.
* Participants with active interstitial lung disease (ILD)/pneumonitis or history of ILD/ pneumonitis requiring steroids.
* Prior treatment with BMS-986205 or any other IDO1 inhibitors.
* Quantitative or qualitative G6PD assay results suggesting underlying G6PD deficiency.
* Blood methemoglobin > upper limit of normal (ULN), assessed in an arterial or venous blood sample or by co-oximetry.
* History or presence of hypersensitivity or idiosyncratic reaction to methylene blue.
* History of allergy or hypersensitivity to any study treatment components, specifically to that of BMS-986205.
* Any concurrent malignancies; exceptions include- basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer or in situ cervical cancer that has undergone potentially curative therapy. Patients with a history of other prior malignancy must have been treated with curative intent and must have remained disease-free for 2 years post-diagnosis.
* Any diagnosis of immunodeficiency or receiving systemic steroid therapy (> 10 mg daily prednisone equivalents) or any other form of immunosuppressive therapy within 14 days of initiation of therapy.
* Patients that have an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids (> 10 mg daily prednisone equivalents) or immunosuppressive agents. Subjects with vitiligo, type I diabetes mellitus, or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study.
* Patients must not be receiving any other investigational agents.
* Patients with uncontrolled intercurrent illnesses including, but not limited to an active infection requiring systemic therapy or a known psychiatric or substance abuse disorder(s) that would interfere with cooperation with the requirements of the trial.
* Patients must not be pregnant or breastfeeding.
* Patients with a known human immunodeficiency virus infection (HIV 1/2 antibodies) or acquired immunodeficiency syndrome (HIV/AIDS), active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected).
* Patients with any evidence of current interstitial lung disease (ILD) or pneumonitis.
* Patients with prior history of ILD or non-infectious pneumonitis that required steroids.
* Patients who have received a live vaccine within 30 days of the planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response | At 5 weeks
  Will be assessed by computed tomography (CT) or magnetic resonance imaging (MRI) scans. The proportions of the primary endpoint in the two treatment groups will be compared at 25% significance level using a two-sided test in proportions. Will re-analyze the primary endpoints using a combined patients collection. Historical controls of patients who received nivolumab alone for 4 weeks in previous window of opportunity trial (CA209-9A7) will be included in the control group. Patients' demographic as well as pre-treatment clinical measurements will be compared between the combined control group versus the treatment group to ensure the homogeneity of the two groups. A multi-variable logistic regression model will be used in the statistical analysis, if any difference in the demographic and clinical predictors between treatment groups is detected. Otherwise, the proportions of the primary endpoint in the two treatment groups will be compared at 5% significance level using a two-sided test.

SECONDARY OUTCOMES:
Objective pathologic response at time of surgery | At time of surgery
  If there is at least one significant difference between groups among the primary outcomes, the two randomization arms will be compared with respect to each secondary outcome using two-sample t-tests. P-values for comparisons of changes in secondary outcomes will be adjusted using the method of Benjamini and Hochberg to control the false discovery rate (FDR) among the secondary outcomes at 5%.
Change in immune cell polarization (Th1/Th2; M1/M2) in peripheral blood and tumor specimens | Baseline up to 12 months
  Will be analyzed and compared using multiplex cytokine analysis collected before and after exposure to nivolumab +/- IDO1 inhibitor BMS-986205 (BMS986205). If there is at least one significant difference between groups among the primary outcomes, the two randomization arms will be compared with respect to each secondary outcome using two-sample t-tests. P-values for comparisons of changes in secondary outcomes will be adjusted using the method of Benjamini and Hochberg to control the FDR among the secondary outcomes at 5%.
Change in inflammatory markers | Baseline up to 12 months
  These include soluble (s)CD40 ligand (L), EGF, eotaxin, FGF-2, Flt-3 ligand, fractalkine, granulocyte colony-stimulating factor (G-CSF), granulocyte colony-macrophage (GM)-CSF, GRO, IFN-alpha2, IL-1alpha, IL-1beta, IL-1ra, IL-3, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-12 (p40), IL-13, IL-15, IL-17A, IP-10, MCP-1, MCP-3, MDC (CCL22), MIP-1alpha, MIP-1beta, PDGF-AA, PDGF-AB/BB, RANTES, TGF-alpha, TNF-alpha, VEGF. If there is at least one significant difference between groups among the primary outcomes, the two randomization arms will be compared with respect to each secondary outcome using two-sample t-tests. P-values for comparisons of changes in secondary outcomes will be adjusted using the method of Benjamini and Hochberg to control the FDR among the secondary outcomes at 5%
Change in prevalence of intratumoral immune cell populations (effector T cells [Teff], regulatory T cells [Treg], and tumor-associated macrophages [TAM] in patients treated with Nivolumab and BMS986205 as compared to patients treated with Nivolumab alone | Baseline up to 12 months
  Assessed by immunohistochemistry (IHC). If there is at least one significant difference between groups among the primary outcomes, the two randomization arms will be compared with respect to each secondary outcome using two-sample t-tests. P-values for comparisons of changes in secondary outcomes will be adjusted using the method of Benjamini and Hochberg to control the FDR among the secondary outcomes at 5%.
Localization of immune cells within the tumor | Up to 12 months
  Will be analyzed using confocal microscopy.
Multiplex colocalization of resident immune cells | Up to 12 months
  Will utilize 5-6 markers per section.
Kynurenine levels (blood and tumor) | Up to 12 months
  Measured with commercial quantitative enzyme-linked immunosorbent assay (ELISA) kits. If there is at least one significant difference between groups among the primary outcomes, the two randomization arms will be compared with respect to each secondary outcome using two-sample t-tests. P-values for comparisons of changes in secondary outcomes will be adjusted using the method of Benjamini and Hochberg to control the FDR among the secondary outcomes at 5%.
Intratumoral immune cell populations, immune polarization data, exosome composition, and exosome function in human papilloma virus (HPV) + and HPV- tumors | Up to 12 months
  Baseline IHC staining for P16 will be performed as a surrogate for HPV status. If there is at least one significant difference between groups among the primary outcomes, the two randomization arms will be compared with respect to each secondary outcome using two-sample t-tests. P-values for comparisons of changes in secondary outcomes will be adjusted using the method of Benjamini and Hochberg to control the FDR among the secondary outcomes at 5%.
Intratumoral immune cell populations, immune polarization data, exosome composition, and exosome function relative to PD-L1 expression levels | Up to 12 months
  Assessed by IHC. If there is at least one significant difference between groups among the primary outcomes, the two randomization arms will be compared with respect to each secondary outcome using two-sample t-tests. P-values for comparisons of changes in secondary outcomes will be adjusted using the method of Benjamini and Hochberg to control the FDR among the secondary outcomes at 5%.
Incidence of adverse events | Up to 100 days
  Will be graded by Common Terminology Criteria for Adverse Events version 5.0. Safety outcomes will be summarized overall and by treatment arm.

OTHER OUTCOMES:
Intratumoral T-cell receptor (TCR) repertoire and diversity | Up to 12 months
  Assesses with next generation sequencing.
Change in exosome abundance and composition in the peripheral blood of patients both before and after exposure to both nivolumab and BMS986205 and nivolumab alone | Baseline up to 12 months
  Will be compared between treatment arms using two-sample t-tests.
Rates of wound dehiscence, postop wound infection (requiring antibiotics), and fistula formation | Up to 12 months
  Will be summarized by treatment arm and compared using Fisher's exact test.
Changes in tumor volume and rates of radiographic response | Baseline up to 12 months
  Will be summarized by treatment arm and compared using two-sample t-tests or Fisher's exact test, as appropriate.
Patient-reported outcomes | Up to 12 months
  Data will be collected and correlated to both immune cell composition and polarization and tumor radiographic response using scores from Patient Health Questionnaire (PHQ)2/9, Functional Assessment of Cancer Therapy- General (FACT-G), and FACT-head and neck (HN). Will conduct descriptive statistics and will summarize variable of interest using standard statistics such as frequency tables, means, and standard deviations. All measures will be evaluated for reliability and factor analyses will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Luginbuhl, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (2):
- United States (2):
  - Ohio State University, Columbus, Ohio
  - Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania

REFERENCES:
- See also: Sidney Kimmel Cancer Center — https://www.jeffersonhealth.org/clinical-specialties/cancer
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/